CLINICAL TRIAL: NCT02259985
Title: Investigation of the Effects of Food on the Bioavailability and Pharmacokinetic Profile of Itasetron After a Single Oral Dose of 1 mg in Healthy Male Subjects (3-way Cross-over)
Brief Title: Effects of Food on the Bioavailability and Pharmacokinetic Profile of Itasetron After a Single Oral Dose in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 208.629
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — itasetron

ARMS (3):
- Itasetron tablet fed (Experimental)
  Interventions: Drug: Itasetron tablet; Other: high fat breakfast
- Itasetron tablet fasted (Active Comparator)
  Interventions: Drug: Itasetron tablet
- Itasetron infusion fasted (Active Comparator)
  Interventions: Drug: Itasetron infusion

INTERVENTIONS:
Drug: Itasetron tablet
  Arms: Itasetron tablet fasted; Itasetron tablet fed
Drug: Itasetron infusion
  Arms: Itasetron infusion fasted
Other: high fat breakfast
  Arms: Itasetron tablet fed

SUMMARY:
food interaction, pharmacokinetics, safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* all participants in the study will range from 21 to 50 years of age and be within +- 20% of their normal weight (Broca-index)
* written informed consent in accordance with Good Clinical Practica and local legislation

Exclusion Criteria:

* Subjects will be excluded from the study if the results of the medical examination or laboratory tests are judged by the investigator to differ significantly from normal clinical values
* Subjects with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Subjects with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* Subjects with known history of orthostatic hypotension, fainting spells or blackouts
* Subjects with chronic or relevant acute infections
* Subjects with history of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Subjects who have taken a drug with a long half-life (>= 24 hours) within one month before enrolment in the study
* Subjects who received any other drugs which might influence the results of the trial during the week previous the start of the study
* Subjects who have participated in another study with an investigational drug within the last 2 months preceding this study
* Subjects who are unable to refrain from smoking on study days
* Subjects who smoke more than 10 cigarettes (or 3 cigars or pipes) per day
* Subjects who drink more than 60 g of alcohol per day
* Subjects who are dependent on drugs
* Subjects who have donated blood (>= 100 ml) within the last 4 weeks
* Subjects who participated in excessive physical activities (e.g. competitive sports) within the last week before the study

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 1998-03; Primary Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve from zero to infinity (AUC0-inf) | up to 48 hours after drug administration
Maximum concentration of drug in plasma | up to 48 hours after drug administration
Time to maximum concentration (tmax) | up to 48 hours after drug administration

SECONDARY OUTCOMES:
Area under the concentration time curve from zero to to the time of last data point above limit of quantitation (AUC0-tlast) | up to 48 hours after drug administration
Cmax/AUC ratio | up to 48 hours after drug administration
Mean residence time in the body (MRTtot) | up to 48 hours after drug administration
Elimination half-life (t1/2) | up to 48 hours after drug administration
Apparent volume of distribution during the terminal phase λz (Vz) | up to 48 hours after drug administration
Total clearance from plasma (CLtot) | up to 48 hours after drug administration
Apparent volume of distribution after intravascular dose at steady state (Vss) | up to 48 hours after drug administration
Number of participants with clinically significant findings in vital signs | up to 8 days after last drug administration
  blood pressure, pulse rate
Number of participants with clinically significant findings in ECG | up to 8 days after last drug administration
Number of participants with clinically significant findings in laboratory tests | up to 8 days after last drug administration
Number of participants with adverse events | up to 8 days after last drug administration